CLINICAL TRIAL: NCT02770157
Title: Phase III Clinical Trial for Assessment of Efficacy and Safety of DA-3002 (Recombinant Human Growth Hormone) in Short Children Born Small for Gestational Age.
Brief Title: Efficacy and Safety of DA-3002 in Short Children Borns SGA.
Acronym: SGA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA3002_SGA_III
Record Dates: First submitted 2016-05-10; First posted 2016-05-12 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Infant, Small for Gestational Age
MeSH Terms: interventions — Human Growth Hormone

ARMS (3):
- DA-3002 (Experimental): 1.44 IU (0.48mg)/kg/week of DA-3002 is injected for 52 weeks by changing injecting areas(six or seven times per week).
  Interventions: Drug: DA-3002
- Genotropin® (Active Comparator): 1.44 IU (0.48mg)/kg/week of Genotropin is injected for 52 weeks by changing injecting areas(six or seven times per week).
  Interventions: Drug: Genotropin®
- Non-treatment control group (Other): After no treatment for 26 weeks, 1.44 IU (0.48mg)/kg/week of DA-3002 is injected for 52 weeks by changing injecting areas(six or seven times per week).
  Interventions: Drug: DA-3002

INTERVENTIONS:
Drug: DA-3002
  Arms: DA-3002; Non-treatment control group
Drug: Genotropin®
  Arms: Genotropin®

SUMMARY:
A study demonstrates the non-inferiority of DA-3002 when compared with Genotropin® in short children born small for gestational age.

ELIGIBILITY:
Inclusion Criteria:

* Chronological Age ≥ 4
* Before the adolescence, Tuner stage I (breast)
* Height <3rd percentile for age
* Normal thyroid function

Exclusion Criteria:

* Growth hormone was administered for 12 months or longer in the past
* Treated with estrogen or adrenal androgens for 12 months or longer in the past
* Malignancy, CNS Trauma, Psychiatric Disorder
* endocrine and/or metabolic disorders
* growth failure caused by other disorders

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2016-02-26 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Annualized height velocity(cm/year) after 52 weeks. | 52 weeks
  Height velocity calculated with height measured at Baseline and after 52 weeks was converted to annual growth rate.

SECONDARY OUTCOMES:
Annualized height velocity(cm/year) after 26 weeks. | 26 weeks
  Height velocity calculated with height measured at Baseline and after 26 weeks was converted to annual growth rate.
Changes in height standard deviation score after 52 weeks | 52 weeks
Changes in bone maturation(changes in bone ages/changes in chronological age) after 52 weeks | 52 weeks
Changes in IGF-1 after 52 weeks | 52 weeks
Changes in IGFBP-3 after 52 weeks | 52 weeks

OTHER OUTCOMES:
Changes in anti-growth hormone antibody | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dong kyu Jin, M.D., Ph.D., Principal Investigator — Seoul Samsung Medical center.; Byung Kyu Suh, M.D., Ph.D., Principal Investigator — Seoul St. Mary's Hospital, The Catholic University of Korea; Cheol Woo Ko, M.D., Ph.D., Principal Investigator — Kyungpook National University Hospital; Kee Hyoung Lee, M.D., Ph.D., Principal Investigator — Korea University Anam Hospital; Han Wook Yoo, M.D., Ph.D., Principal Investigator — Asan Medical Center; Choong Ho Shin, M.D., Ph.D., Principal Investigator — Seoul National University Hospital; Jin Soon Hwang, M.D., Ph.D., Principal Investigator — Aju University Hospital; Ho Seong Kim, M.D., Ph.D., Principal Investigator — Severance Children's Hospital Yonsei University; Woo Young Jeong, M.D., Ph.D., Principal Investigator — Pusan University Hospital; Chang Jong Kim, M.D., Ph.D., Principal Investigator — Chonnam National University Hospital; Heon Suk Han, M.D., Ph.D., Principal Investigator — Chungbuk National University Hospital
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim SJ, Kim MS, Cho SY, Suh BK, Ko CW, Lee KH, Yoo HW, Shin CH, Hwang JS, Kim HS, Chung WY, Kim CJ, Han HS, Jin DK. Efficacy and safety of the recombinant human growth hormone in short children born small for gestational age: A randomized, multicentre, comparative phase III trial. Medicine (Baltimore). 2021 Jul 30;100(30):e26711. doi: 10.1097/MD.0000000000026711. PMID 34397702